CLINICAL TRIAL: NCT01158664
Title: A Prospective Multicenter Randomized Controlled Clinical Study on Conical Southern Implants With Different Thread Pitch
Brief Title: What is the Influence of a Different Thread Pitch Design on Bone Remodelling Around Conical Southern Oral Implants?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009/649
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Dental Implants
Keywords: dental implants; different tread pitch design

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.6 mm tread pitch implant (Experimental)
  Interventions: Device: 0.6 mm tread pitch implant
- 0.1 mm tread pitch implant (Experimental)
  Interventions: Device: 0.1 mm tread pitch implant

INTERVENTIONS:
Device: 0.6 mm tread pitch implant — 0.6 mm tread pitch implant will be used
  Arms: 0.6 mm tread pitch implant
Device: 0.1 mm tread pitch implant — 0.1 mm tread pitch implant will be used
  Arms: 0.1 mm tread pitch implant

SUMMARY:
Patients who need more than 2 dental implants will be treated by the same implant type (conical 4mm diameter IBT Southern implants) but with different thread pitch design (0,6mm en 1,0mm type). In a 3 year clinical follow up period, the bone remodelling on X-rays is registered around these implants. The role of the thread pitch design will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Periodontally-healthy or periodontally-treated patients
* Smokers are included
* All types of prosthetic indications are accepted but 2 IBT type implants with different threads have to be placed in one patient on the same day. Implants can be connected or not connected in the same jaw.

Exclusion Criteria:

* All other contra indications for implant surgery
* Guided bone regeneration or use of any substitutes
* No implantation in regenerated or augmented bone
* No immediate loading cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To document the outcome of bone remodeling around IBT implants | 3 years after implantation

SECONDARY OUTCOMES:
To clinically and radiographically document the placement of both IBT implant thread types in the same patient | over 2 years
3. Outcome differences will be detected per implant center, per treated area in the mouth, per case of prosthetic rehabilitation | over 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hugo De Bruyn, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website of University Hospital Ghent, Belgium — http://www.uzgent.be